CLINICAL TRIAL: NCT00890097
Title: The Safety and Efficacy of AL-8309B Ophthalmic Solution for the Treatment of Geographic Atrophy (GA) Secondary to Age-Related Macular Degeneration (AMD)
Brief Title: Geographic Atrophy Treatment Evaluation
Acronym: GATE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Treatment ineffective
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-08-36
Record Dates: First submitted 2009-04-27; First posted 2009-04-29 (Estimated); Results first posted 2014-07-03 (Estimated); Last update posted 2014-07-03 (Estimated); Status verified 2014-06

CONDITIONS: Geographic Atrophy; Age-Related Macular Degeneration
Keywords: Geographic Atrophy; GA; Age-Related Macular Degeneration; AMD
MeSH Terms: conditions — Geographic Atrophy; Macular Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- AL-8309B 1.0% (Experimental): AL-8309B 1.0% Ophthalmic Solution, 1 drop in each eye twice daily for 30 months, up to a maximum of 36 months
  Interventions: Drug: AL-8309B Ophthalmic Solution
- AL-8309B 1.75% (Experimental): AL-8309B 1.75% Ophthalmic Solution, 1 drop in each eye twice daily, for 30 months up to a maximum of 36 months
  Interventions: Drug: AL-8309B Ophthalmic Solution
- Vehicle (Placebo Comparator): AL-8309B Vehicle, 1 drop in each eye twice daily, for 30 months up to a maximum of 36 months
  Interventions: Drug: AL-8309B Vehicle

INTERVENTIONS:
Drug: AL-8309B Ophthalmic Solution
  Arms: AL-8309B 1.0%; AL-8309B 1.75%
Drug: AL-8309B Vehicle — Inactive ingredients used as placebo comparator
  Arms: Vehicle

SUMMARY:
The purpose of this study was to evaluate the safety and efficacy of AL-8309B Ophthalmic Solution versus Vehicle administered as a topical ocular drop for the treatment for geographic atrophy (GA) secondary to age-related macular degeneration (AMD).

ELIGIBILITY:
Inclusion Criteria:

* Willing to give written informed consent, make required study visits, and follow instructions.
* Able to administer eye drops or have a caretaker to administer the eye drops.
* Study eye: Atrophy secondary to age-related macular degeneration, best corrected visual acuity (BCVA) of 35 letters (20/200 Snellen equivalent) or better, clear ocular media, and adequate pupillary dilation.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Pregnant, nursing, or not using adequate contraception.
* Ocular disease in the study eye, other than non-exudative AMD.
* History of cataract surgery in either eye within the past 3 months of screening.
* History or evidence of serious ocular trauma or intraocular surgery in either eye within the past 6 months of screening.
* Any medical condition that would make participation in the trial or adherence to the study schedule difficult or unlikely.
* Participation in an investigational drug or device study within 30 days of screening.
* Other protocol-defined exclusion criteria may apply.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 772 (Actual)
Dates: Start 2009-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sally Scheib, Sr. Clinical Lead, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 48 study centers located in 14 countries.
Pre-assignment Details: This reporting group includes all enrolled subjects (772). A subject was considered enrolled if they met all of the inclusion criteria and none of the exclusion criteria.
Period: Overall Study
Arm/Group | AL-8309B 1.0% | AL-8309B 1.75% | Vehicle
Started | 252 | 259 | 261
Completed | 184 | 173 | 184
Not Completed | 68 | 86 | 77
Not completed — Adverse Event | 21 | 32 | 28
Not completed — Decision Unrelated to an Adverse Event | 15 | 12 | 17
Not completed — Withdrew Consent | 9 | 6 | 9
Not completed — Lost to Follow-up | 5 | 5 | 5
Not completed — Noncompliance | 0 | 4 | 4
Not completed — Sponsor Decision | 7 | 11 | 7
Not completed — Did not attend final visit | 2 | 3 | 0
Not completed — Subject Decision | 3 | 2 | 6
Not completed — Randomization Error | 2 | 0 | 0
Not completed — Failed inclusion criteria | 3 | 4 | 0
Not completed — Transportation | 0 | 2 | 0
Not completed — Subject Moved | 0 | 4 | 0
Not completed — Protocol Deviation | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: This analysis population includes all enrolled subjects (772).
Groups:
- Total: Total of all reporting groups
Arm/Group | AL-8309B 1.0% | AL-8309B 1.75% | Vehicle | Total
Number analyzed (Participants) | 252 | 259 | 261 | 772
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.9 (8.0) | 78.3 (7.7) | 78.8 (7.1) | 78.3 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130 | 162 | 147 | 439
  Male | 122 | 97 | 114 | 333
Region of Enrollment [Number; unit: participants]
  United States | 111 | 112 | 116 | 339
  France | 28 | 27 | 29 | 84
  Switzerland | 21 | 21 | 21 | 63
  Germany | 18 | 20 | 19 | 57
  Australia | 16 | 18 | 16 | 50
  Israel | 13 | 15 | 15 | 43
  Italy | 12 | 15 | 14 | 41
  Austria | 13 | 13 | 14 | 40
  Belgium | 7 | 6 | 6 | 19
  United Kingdom | 4 | 3 | 3 | 10
  Ireland | 3 | 3 | 3 | 9
  Japan | 3 | 2 | 3 | 8
  Portugal | 2 | 3 | 2 | 7
  Canada | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean Annualized Lesion Enlargement Rate From Baseline as Assessed With Fundus Autofluorescence Imaging
Description: The size of the retinal lesion was measured using the Heidelberg Retinal Angiography system at Baseline, Month 6, Month 12, Month 15, Month 18, Month 24, and Month 30. Images were collected in both eyes; however, one eye from each subject was chosen as the study eye, and only data for the study eye were used for the efficacy analysis. Results were estimated from a longitudinal random effects regression model. A greater lesion growth rate may indicate a faster progression of the disease.
Time Frame: Baseline, up to Month 30
Population: This analysis population included all treated subjects. A subject was considered treated if they had a first or last dosing date in the database.
Measure: Mean (95% Confidence Interval); unit: square millimeters per year
Arm/Group | AL-8309B 1.0% | AL-8309B 1.75% | Vehicle
Number analyzed (Participants) | 250 | 258 | 260
square millimeters per year | 1.725 [1.595 to 1.855] | 1.758 [1.626 to 1.890] | 1.707 [1.585 to 1.830]

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study (3 years, 2 month). Adverse events were obtained as solicited comments from the study subjects and as observations by the study Investigator as outlined in the study protocol.
Description: This analysis population includes all treated subjects (768).
Arm/Group | AL-8309B 1.0% | AL-8309B 1.75% | Vehicle
Serious Adverse Events (participants affected / at risk) | 86/250 | 96/258 | 85/260
Other Adverse Events (participants affected / at risk) | 207/250 | 212/258 | 207/260
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AL-8309B 1.0% (N=250) | AL-8309B 1.75% (N=258) | Vehicle (N=260)
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 1 | 0
Angina pectoris (Cardiac disorders) | 4 | 3 | 1
Angina unstable (Cardiac disorders) | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 1
Arrhythmia supraventricular (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 4 | 3 | 5
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 1
Bundle branch block (Cardiac disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0
Cardiac disorder (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 2 | 4 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 4 | 3 | 1
Coronary artery disease (Cardiac disorders) | 0 | 2 | 1
Coronary artery occlusion (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 4 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 1 | 0
Sinus arrhythmia (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 2
Choledochal cyst (Congenital, familial and genetic disorders) | 0 | 1 | 0
Goitre (Endocrine disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 1
Macular oedema (Eye disorders) | 0 | 1 | 0
Retinal artery occlusion (Eye disorders) | 0 | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 1 | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 | 1 | 0
Intussusception (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 2
Chest discomfort (General disorders) | 0 | 0 | 1
Chest pain (General disorders) | 3 | 1 | 0
Death (General disorders) | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 0 | 1
Impaired healing (General disorders) | 0 | 0 | 1
Inflammation (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 1
Pain (General disorders) | 2 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 0
Biliary tract disorder (Hepatobiliary disorders) | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Cirrhosis alcoholic (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1 | 0
Anaphylactic shock (Immune system disorders) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 1
Dacryocystitis (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 4 | 0 | 0
Echinococciasis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 2
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0
Labyrinthitis (Infections and infestations) | 0 | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 0 | 1
Localised infection (Infections and infestations) | 1 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 2
Lung infection (Infections and infestations) | 0 | 0 | 1
Pancreatic abscess (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 3 | 9 | 5
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 3 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 3 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1
Injury (Injury, poisoning and procedural complications) | 16 | 14 | 15
Intraocular lens dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 2 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 1
Arthroscopy (Investigations) | 1 | 0 | 0
Catheterisation cardiac (Investigations) | 2 | 1 | 1
Endoscopy (Investigations) | 1 | 0 | 0
Investigation (Investigations) | 0 | 0 | 2
Oxygen saturation decreased (Investigations) | 0 | 0 | 1
Renal function test abnormal (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 5 | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cardiac valve fibroelastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hepatic neoplasm malignant non-resectable (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung adenocarcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to abdominal cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 0
Pancreatic carcinoma non-resectable (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Ureteric cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 0
Cerebral artery occlusion (Nervous system disorders) | 0 | 1 | 0
Cerebral haematoma (Nervous system disorders) | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 3 | 4 | 3
Convulsion (Nervous system disorders) | 1 | 0 | 0
Dementia (Nervous system disorders) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 0 | 1
Extrapyramidal disorder (Nervous system disorders) | 0 | 1 | 0
Grand mal convulsion (Nervous system disorders) | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 2
Headache (Nervous system disorders) | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 2 | 0 | 0
Nerve compression (Nervous system disorders) | 0 | 1 | 0
Parkinson's disease (Nervous system disorders) | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 2 | 2
Syringomyelia (Nervous system disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 4 | 2 | 2
Confusional state (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0
Depression suicidal (Psychiatric disorders) | 0 | 1 | 0
Disorientation (Psychiatric disorders) | 0 | 1 | 1
Hallucination, visual (Psychiatric disorders) | 0 | 0 | 1
Major depression (Psychiatric disorders) | 0 | 1 | 1
Mental status changes (Psychiatric disorders) | 1 | 1 | 0
Schizophrenia (Psychiatric disorders) | 1 | 0 | 0
Bladder disorder (Renal and urinary disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Pelvi-ureteric obstruction (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 1 | 1
Renal failure chronic (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 3 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0
Prostatomegaly (Reproductive system and breast disorders) | 1 | 1 | 0
Vaginal fistula (Reproductive system and breast disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Angioplasty (Surgical and medical procedures) | 0 | 1 | 0
Aortic aneurysm repair (Surgical and medical procedures) | 0 | 1 | 0
Aortic valve repair (Surgical and medical procedures) | 0 | 0 | 1
Aortic valve replacement (Surgical and medical procedures) | 0 | 1 | 0
Appendicectomy (Surgical and medical procedures) | 0 | 1 | 0
Bunion operation (Surgical and medical procedures) | 0 | 0 | 1
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 | 0 | 1
Cardioversion (Surgical and medical procedures) | 0 | 0 | 1
Haemorrhoid operation (Surgical and medical procedures) | 1 | 0 | 0
Hip arthroplasty (Surgical and medical procedures) | 0 | 2 | 1
Hip surgery (Surgical and medical procedures) | 0 | 0 | 1
Inguinal hernia repair (Surgical and medical procedures) | 0 | 0 | 1
Intraocular lens implant (Surgical and medical procedures) | 1 | 0 | 0
Intrathecal pump insertion (Surgical and medical procedures) | 1 | 0 | 0
Joint arthroplasty (Surgical and medical procedures) | 0 | 0 | 1
Keratoplasty (Surgical and medical procedures) | 0 | 1 | 0
Knee arthroplasty (Surgical and medical procedures) | 2 | 1 | 0
Knee operation (Surgical and medical procedures) | 0 | 1 | 1
Malignant tumour excision (Surgical and medical procedures) | 0 | 1 | 0
Radiotherapy to eye (Surgical and medical procedures) | 1 | 0 | 0
Salivary gland operation (Surgical and medical procedures) | 0 | 1 | 0
Scoliosis surgery (Surgical and medical procedures) | 1 | 0 | 0
Spinal operation (Surgical and medical procedures) | 0 | 0 | 1
Vasodilation procedure (Surgical and medical procedures) | 0 | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 1 | 0
Aortic stenosis (Vascular disorders) | 1 | 1 | 0
Arterial occlusive disease (Vascular disorders) | 0 | 1 | 1
Circulatory collapse (Vascular disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 2 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 1
Temporal arteritis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AL-8309B 1.0% (N=250) | AL-8309B 1.75% (N=258) | Vehicle (N=260)
Blepharitis (Eye disorders) | 15 | 19 | 7
Cataract (Eye disorders) | 30 | 23 | 23
Choroidal neovascularisation (Eye disorders) | 20 | 20 | 16
Eye irritation (Eye disorders) | 20 | 27 | 9
Eye pain (Eye disorders) | 16 | 21 | 11
Lacrimation increased (Eye disorders) | 8 | 15 | 3
Macular degeneration (Eye disorders) | 18 | 20 | 14
Retinal haemorrhage (Eye disorders) | 14 | 16 | 21
Visual acuity reduced (Eye disorders) | 101 | 107 | 109
Constipation (Gastrointestinal disorders) | 13 | 4 | 13
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 15 | 11 | 9
Nausea (Gastrointestinal disorders) | 15 | 8 | 8
Oedema peripheral (General disorders) | 14 | 4 | 11
Bronchitis (Infections and infestations) | 15 | 21 | 28
Influenza (Infections and infestations) | 7 | 8 | 14
Nasopharyngitis (Infections and infestations) | 19 | 19 | 22
Urinary tract infection (Infections and infestations) | 20 | 28 | 19
Injury (Injury, poisoning and procedural complications) | 34 | 38 | 31
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 15 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 12 | 17
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 14 | 21 | 12
Headache (Nervous system disorders) | 19 | 15 | 9
Depression (Psychiatric disorders) | 10 | 9 | 18
Hypertension (Vascular disorders) | 24 | 30 | 36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.